CLINICAL TRIAL: NCT04536402
Title: A Multi-centre, Prospective, Observational Post-Authorization Safety Study to Evaluate the Safety Profile of Budesonide/Glycopyrrolate/Formoterol MDI in Chinese Patients With COPD in Routine Clinical Practice
Brief Title: Evaluate the Safety Profile of BGF MDI in Chinese Patients With COPD in Routine Clinical Practice
Acronym: TORES
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00016
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — no sample collect in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational, multicenter, prospective, single arm study. The objective of this study is to evaluate the safety of Breztri® Aerosphere® in Chinese patients with COPD in real world clinical practice. The study will enrol approximately 3,050 subjects from about 42 sites around China and followed up for 12 weeks.

DETAILED DESCRIPTION:
This study is an observational, multicenter, prospective, single arm study. 3,050 subjects who have been prescribed and have planned to take at least one inhalation of BGF MDI will be enrolled into the study

This is an observational study. BGF MDI treatment will be studied through non-interventional approach. It will be carried out under routine clinical practice and the start or end of BGF MDI and other concomitant treatment will be determined by subjects' treating physicians.

Eligible subjects will be consecutively enrolled in this study at the time they routinely visit their physician and consent to participate in the study. After enrolled successfully, baseline variables will be collected at V1. Subjects will be followed up every 4 weeks after baseline for a total duration of 12 weeks or until study discontinuation, whichever occurs first. V1 and V2 will be followed up by on-site visit and V3 and V4 will be followed up by telephone call visit. For subjects who remain on study drug throughout the study (i.e., complete 4 Visits), a follow up telephone call will be performed at 14 days after the last visit to collect safety information. For subjects who has an Early Discontinuation, 14 days follow up is needed for AE collecting after the discontinuation. For subjects who had been hospitalized during the first 4 weeks of follow-up due to one or more acute exacerbations of COPD, a follow up telephone call will be performed at 28 days after the last visit to collect safety information.

The subjects will be recruited from qualified hospitals. Safety and effectiveness data will be collected following enrollment in the study. Medical records, PROs (COPD Assessment Test [CAT], St. George's Respiratory Questionnaire [SGRQ], Aerosphere Delivery Technology Metered Dose Inhaler Preference Questionnaire [AMPQ], Patient Global Impression of Change [PGIC]) will be the data source in this study.

Primary endpoint will be the incidence of AEs and SAEs in purpose of monitoring the safety profile of BGF MDI.

ELIGIBILITY:
Inclusion Criteria:

* Give their signed written informed consent to participate
* Age: 18 and above
* Chinese, Female or male
* Patient with diagnosis of COPD as defined by clinicians
* Subjects who have been prescribed and have planned to take at least one inhalation of Budesonide/Glycopyrrolate/Formoterol MDI based on physician's decision.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be able to enter the study：

* Subjects who are currently involved in any other interventional studies.
* Drug Allergy: Subjects who have a history of hypersensitivity to formoterol or any other β2-agonists, budesonide or any other corticosteroid components, glycopyrronium or other muscarinic anticholinergics, or any component of the MDI.
* Subjects who received investigational drug treatment within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll 3,050 Chinese COPD patients who have been prescribed and have planned to take at least one inhalation of BGF MDI. The decision to start with BGF MDI treatment is independent of this study.
Sampling Method: Probability Sample
Enrollment: 3520 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence of all AEs /SAEs | 2022-12-30
  To evaluate the safety profile after BGF MDI treatment in Chinese COPD patients

SECONDARY OUTCOMES:
Change from baseline in CAT score | 2022-12-30
  To observe patients' health status after BGF MDI treatment via patient reported outcomes (PROs)
Change from baseline in SGRQ score | 2022-12-30
  To observe patients' health status after BGF MDI treatment via patient reported outcomes (PROs)
ADT MDI preference questionnaire (AMPQ) | 2022-12-30
  To describe patient preference for the Aerosphere Delivery Technology
Patient global impression of change (PGIC) | 2022-12-30
  To observe patients' health status after BGF MDI treatment via patient reported outcomes (PROs)
Mean total COPD cost including the direct and indirect COPD cost | 2022-12-30
  To assess total direct and indirect COPD cost

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, Principal Investigator — Peking Universicy Third Hospital
Locations (29):
- China (29):
  - Research Site, Beijing
  - Research Site, Changzhi
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Chongqing
  - Research Site, Guangyuan
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Haining
  - Research Site, Hangzhou
  - Research Site, Huizhou
  - Research Site, Jiaxing
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Jinzhong
  - Research Site, Mianyang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Taizhou
  - Research Site, Weifang
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xinxiang
  - Research Site, Xinzheng
  - Research Site, Yangquan
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
  - Research Site, Zibo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00016&attachmentIdentifier=f823a1d1-d306-4efa-b8e0-d184b96b1e43&fileName=TORES_CSR_Synopsis_.pdf&versionIdentifier=